CLINICAL TRIAL: NCT03078855
Title: ILyAD (Indolent Lymphoma And Vitamin D) A Phase III Double Blind, Randomized Trial to Evaluate the Effect of Vitamin D on Progression-free Survival in Patients With Low Tumor-burden Indolent Non-Hodgkin Lymphoma Treated With Rituximab
Brief Title: A Study to Evaluate the Effect of Vitamin D on PFS in Indolent Non-Hodgkin's Lymphoma
Acronym: ILyAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonathan Friedberg (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jonathan Friedberg, Director, Wilmot Cancer Institute, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 66593; R01CA214890 (NIH)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Follicular Lymphoma; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma; Mucosal-Associated Lymphoid Tissue Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Vitamin D; Cholecalciferol; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D plus rituximab (Experimental): Rituximab was administered weekly x 4 (intravenous 375 mg/m^2 or subcutaneous equivalent) per institutional standards and vitamin D3, 2000 IU orally once daily. Participants took vitamin D3 until lack of response at week 13, disease progression, or initiation of a new treatment.
  Interventions: Dietary Supplement: Vitamin D; Biological: Rituximab
- Placebo plus rituximab (Placebo Comparator): Rituximab was administered weekly x 4 (intravenous 375 mg/m^2 or subcutaneous equivalent) per institutional standards and placebo orally once daily. Participants took placebo until lack of response at week 13, disease progression, or initiation of a new treatment.
  Interventions: Biological: Rituximab; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — vitamin D3 2,000 IU daily
  Other Names: Cholecalciferol
  Arms: Vitamin D plus rituximab
Biological: Rituximab — Administered weekly x 4
  Other Names: Rituxan
Other: Placebo — methylcellulose
  Arms: Placebo plus rituximab

SUMMARY:
Despite strong evidence suggesting that vitamin D deficiency is associated with undesirable outcomes in patients with numerous cancers, there has never been a thorough study of vitamin D treatment in subjects undergoing treatment for cancer. The purpose of this study is to evaluate whether modification of vitamin D levels in the blood, through supplementation, can improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Each of the following criteria must be met in order for a patient to be considered eligible for registration:

* Biopsy proven (with hematopathology review at one of the participating sites to confirm correct histology in accordance with World Health Organization) indolent lymphoma to include the following diagnoses:

  * Grade 1, 2, or 3a follicular lymphoma
  * Small lymphocytic lymphoma (CLL excluded)
  * Marginal zone lymphoma (nodal or splenic)
  * Mucosal-associated lymphoid tissue
* Measurable disease defined by Lugano criteria
* No prior anti-lymphoma systemic therapy; prior radiation therapy allowed
* Age 18 or over
* Ann Arbor stages II, III or IV
* Patients with follicular lymphoma must have PET FDG-avid lymphoma and fulfill Low tumor burden by Groupe D'Etude des Lymphomes Folliculaires (GELF) criteria:

  * No mass > 7 cm
  * < 3 distinct masses of greater than 3 cm
  * No B symptoms
  * No splenomegaly > 16 cm by computed tomography (CT) scan
  * No risk of vital organ compression
  * No leukemic phase > 5000/µl circulating lymphocytes (except for in patients with splenic marginal zone diagnosis)
  * No cytopenias (platelets < 100,000/µl, hemoglobin < 10 g/dl, or absolute neutrophil count < 1500/µl)

Exclusion Criteria:

The following criteria will prevent inclusion of an inappropriate subject into the trial:

* Osteoporosis requiring prescription treatment
* Known symptomatic primary hyperparathyroidism
* Hypercalcemia defined as above the institutional normal range (corrected for albumin when albumin levels are below normal)
* History of calcium-related kidney stones
* Creatinine > 1.5X above upper limit of normal
* Women who are known to be pregnant or who plan to become pregnant while on rituximab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Friedberg, MD, Principal Investigator — James P. Wilmot Cancer Institute at University of Rochester
Locations (7):
- United States (7):
  - University of Miami, Miami, Florida
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - James P. Wilmot Cancer Institute at University of Rochester Medical Center, Rochester, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests will be considered beginning in December 2024.

REFERENCES:
- [Derived] Friedberg JW, Brady MT, Strawderman M, Kahl BS, Lossos IS, Cohen JB, Reagan PM, Casulo C, Averill BL, Baran A, Sutamtewagul G, Barr PM, Leonard JP, Ashton JM, Strang JG, Vega F, Peterson DR, Nastoupil LJ. Vitamin D in patients with low tumor-burden indolent non-Hodgkin lymphoma treated with rituximab therapy (ILyAD): a randomized, phase 3 clinical trial. EClinicalMedicine. 2024 Nov 27;78:102959. doi: 10.1016/j.eclinm.2024.102959. eCollection 2024 Dec. PMID 39677358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 US academic medical centers between September 2017 and March 2022.
Period: Overall Study
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab
Started | 139 | 72
Completed | 53 | 32
Not Completed | 86 | 40
Not completed — Lack of Efficacy | 62 | 31
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Physician Decision | 3 | 2
Not completed — Second Malignancy | 4 | 0
Not completed — Ineligible | 2 | 0
Not completed — Withdrew before day 1 treatment | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included randomized and eligible participants that received at least one dose of vitamin D or placebo. Five enrolled participants were either ineligible or withdrew before receiving at least one dose of vitamin D or placebo and were excluded from the baseline analysis population.
Groups:
- Vitamin D Plus Rituximab: Rituximab was administered weekly x 4 (intravenous 375 mg/m^2 or subcutaneous equivalent) per institutional standards and vitamin D3, 2000 IU, was taken orally once daily. Participants took vitamin D3 until lack of response at week 13, disease progression, or initiation of a new treatment.
- Placebo Plus Rituximab: Rituximab was administered weekly x 4 (intravenous 375 mg/m^2 or subcutaneous equivalent) per institutional standards and placebo was taken orally once daily. Participants took placebo until lack of response at week 13, disease progression, or initiation of a new treatment.
- Total: Total of all reporting groups
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab | Total
Number analyzed (Participants) | 135 | 71 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 36 | 116
  >=65 years | 55 | 35 | 90
Age, Continuous [Median (Full Range); unit: years] | 62 [30 to 81] | 64 [39 to 81] | 62 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 40 | 118
  Male | 57 | 31 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 123 | 63 | 186
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 120 | 62 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 135 | 71 | 206

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival
Description: Event free survival (EFS) was defined as the time from randomization to lack of response at week 13, initiation of a new treatment, disease progression defined by Lugano criteria, or death, right-censored by time of last follow-up. Per Lugano criteria, progression is defined as a new FDG-avid lesion or an increase in intensity from baseline, an increase by >= 50% in lesion diameters, a new lymph node > 1.5 cm in any axis or a new extranodal site > 1.0 cm.
Time Frame: 3 years
Population: The analysis population included randomized and eligible participants that received at least one dose of vitamin D or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab
Number analyzed (Participants) | 135 | 71
Percentage of Participants | 47.7 [39.0 to 58.4] | 49.5 [37.6 to 65.0]
Statistical Analysis 1: Comparison: Vitamin D Plus Rituximab vs Placebo Plus Rituximab; Test type: Superiority; p = 0.26, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.83 to 1.98] — The EFS hazard ratio was adjusted for enrolling site, continuous age at randomization, and (via stratification) 3 randomization strata: non-follicular histology, follicular (FL) with low/intermediate FLIPI score and FL with high FLIPI score

2. Secondary Outcome: All-Cause Mortality
Description: Number of participants who died from any cause between day 1 of treatment and the time of last follow-up.
Time Frame: Participants were followed for survival beginning on day 1 of treatment until study closure with a maximum follow-up of 64 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab
Number analyzed (Participants) | 135 | 71
Participants | 4 | 3

3. Secondary Outcome: Number of Participants With Treatment Response at 13 Weeks
Description: Participants had imaging performed at week 13 to assess response to treatment. A response was defined as partial (PR) or complete response (CR) according to Lugano criteria. Per Lugano criteria for target lesions: PR includes reduced metabolic uptake or a ≥ 50% decrease in the sum of the products of the diameters compared to baseline. CR includes metabolic score of 1, 2 or 3 (out of 5) with or without residual mass or regression of target lesions to ≤ 1.5 cm in the longest dimension.
Time Frame: 13 Weeks from the start of treatment
Population: The analysis population included randomized and eligible participants that received at least one dose of vitamin D or placebo and were evaluated for treatment response at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab
Number analyzed (Participants) | 135 | 70
Participants | 113 | 59

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were evaluated beginning on day 1 of treatment through 30 days after the last dose of vitamin D or placebo, up to 37 months. All-cause mortality was evaluated beginning on day 1 of treatment until study closure with a maximum follow-up of 64 months.
Description: Adverse events were collected through chart review and participant solicitation.
Arm/Group | Vitamin D Plus Rituximab | Placebo Plus Rituximab
All-Cause Mortality (participants affected / at risk) | 4/135 | 3/71
Serious Adverse Events (participants affected / at risk) | 16/135 | 9/71
Other Adverse Events (participants affected / at risk) | 111/135 | 54/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D Plus Rituximab (N=135) | Placebo Plus Rituximab (N=71)
Infusion related reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Aortic valve disease (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Other - Hemothorax (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Other - Vision changes (Eye disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Other - COVID19 (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Other - Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Other - Gastric adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Other - Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D Plus Rituximab (N=135) | Placebo Plus Rituximab (N=71)
Chills (General disorders) | 8 | 1
Fatigue (General disorders) | 39 | 19
Fever (General disorders) | 7 | 1
Infusion related reaction (General disorders) | 48 | 22
Injection site reaction (General disorders) | 14 | 8
Abdominal pain (Gastrointestinal disorders) | 11 | 1
Constipation (Gastrointestinal disorders) | 10 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 10 | 6
Other - COVID19 (Infections and infestations) | 12 | 9
Upper respiratory infection (Infections and infestations) | 9 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 7 | 1
Headache (Nervous system disorders) | 18 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 4
Hypertension (Vascular disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT03078855/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03078855/ICF_001.pdf